CLINICAL TRIAL: NCT06043466
Title: Phase I Clinical Study of Chimeric Antigen Receptor T Cells (C-13-60) in the Treatment of Carcinoembryonic Antigen (CEA) Positive Advanced Malignant Solid Tumors
Brief Title: A Clinical Trial Targeting CEA Chimeric Antigen Receptor T (CAR-T) for CEA Positive Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PB06
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Esophagus Cancer; Gastric Cancer; Pancreas Cancer; Non-small Cell Lung Cancer; Breast Cancer; Bile Duct Cancer
Keywords: CAR-T; CEA; CEA-positive advanced/metastatic solid tumors
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 2-10x10^6 cells/kg
  Interventions: Biological: CEA-targeted CAR-T cells

INTERVENTIONS:
Biological: CEA-targeted CAR-T cells — Administration method: intravenous infusion； Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This is a single-arm, open, dose-increasing phase I clinical study to explore the safety, tolerability and pharmacokinetic characteristics of the drug C-13-60 cells, and preliminarily observe the efficacy of the drug in CEA positive late malignant solid tumors, and explore the applicable dose regimen for phase II clinical trials.

DETAILED DESCRIPTION:
According to the sequence principle of low and high dose of C-13-60 cell reinfusion, the dose escalation experiment was carried out successively. Three subjects in each dose group were enrolled first. If DLT did not appear, the decision of whether to enter the next dose group was made according to Safety review committee (SRC) resolution. If there was one case of DLT, then 3 subjects were enrolled one by one, and DLT observation was completed for 28 days after each subject's infusion. If no DLT was found, the next infusion was continued. If DLT was found, the subsequent enrollment of the dose group was terminated, and the experiment was terminated or the dose was reduced according to the dose increasing principle. If > 1 case of DLT occurs, the trial is terminated or the dose is reduced.According to the evaluation of the researchers, the subjects who met the conditions of antisepsis received antisepsis chemotherapy 1-5 to -3 days before the transfusion of C-13-60 cells；

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Patients with advanced malignant solid tumors confirmed by histology or pathology, including colorectal cancer, esophageal cancer, gastric cancer, pancreatic cancer, non-small cell lung cancer, breast cancer, and cholangiocarcinoma;
3. Progression or intolerance occurs after receiving systematic standard therapy according to guidelines,(systemic therapy including but not limited to systemic chemotherapy, molecular targeting, etc.) and is not suitable for surgery or local therapy (including ablative therapy, interventional therapy, and radiation therapy), among which colorectal cancer needs to receive at least third-line therapy failure or intolerance or inapplicability. Esophageal, gastric, non-small cell lung, breast, and cholangiocarcinoma require at least second-line treatment failure or intolerance or inadequacy, and pancreatic cancer require at least first-line treatment failure or intolerance or inadequacy:

   1. Advanced colorectal cancer: progression or intolerance or inadequacy after third-line standard therapy including cetuximab ± Irinotecan/regorafenib /fruquintinib/trifluridine；
   2. Advanced or metastatic esophageal cancer/esophagogastric junction cancer: patients with esophageal cancer who progress or are intolerant or inapplicable after second-line therapy including PD-1 MAB /PD-L1 mab; Patients with esophagogastric junction cancer progressed or were intolerant or inapplicable after second-line therapy including taxane or irinotecan or PD-1 /PD-L1 monoclonal antibody; For HER-2 positive patients, trastuzumab containing system therapy should fail or be intolerable or not applicable;
   3. Advanced/metastatic gastric cancer: the combination of PD-1 MAB /PD-L1 MAB and chemotherapy has been developed or is not tolerated or suitable; For HER-2 positive patients, systemic treatment containing trastuzumab should fail or be intolerable or inapplicable.
   4. Patients with advanced, metastatic, or recurrent non-small cell lung cancer who have received systemic treatment progression or intolerance, including: Patients with positive driver genes (EGFR, ALK, ROS1, BRAF, NTRK, MET, RET) should receive targeted therapy failure or drug resistance (squamous cell carcinoma does not require driver gene testing). In addition, patients with EGFR-positive driver gene who are resistant to first-line EGFR-Tkis and who are positive for EGFR T790M mutations need to be treated with third-generation EGFR-TKI (such as Osimertinib, almonertinib, or furmonertinib) after failure or resistance. For patients with positive ALK fusion and drug resistance after first-line crizotinib treatment, second-line treatment with ceritinib or alectinib should fail or be resistant; Patients with PD-L1 expression (PD-L1 TPS≥1%) should undergo immune checkpoint inhibitor treatment failure or intolerance; In patients with negative driver genes, the disease progresses or becomes intolerable after chemotherapy with platinum-containing regiments-such as Camrelizumab, Pembrolizumab, Tislelizumab, Sintilimab or Atezolizumab combined with pemetrexed
   5. Advanced, metastatic breast cancer: HER-2 positive patients need to have received anti-HER-2 therapy, hormone receptor positive patients need to receive endocrine therapy and other standard treatments have failed or are intolerable or not applicable, and rescue chemotherapy for those who have failed/are intolerable or triple-negative breast cancer (including: Gemcitabine + cisplatin/carboplatin, albumin paclitaxel/other taxoid drugs + cisplatin/carboplatin) fail or are not tolerated or suitable;
   6. Locally advanced or metastatic pancreatic cancer: advanced or intolerant or inappropriate after at least first-line treatment, including: Gemcitabine + albumin-bound paclitaxel/cisplatin/erlotinib/capecitabine/tegafur/Nimotuzumab, or FOLFIRINOX (oxaliplatin + irinotecan +LV+5-FU), or mFOLFIRINOX (oxaliplatin + irinotecan + calcium folinate +5-FU);
   7. Advanced cholangiocarcinoma: progression or intolerance or inapplicability after at least second-line therapy (mFOLFOX); Remarks: Chemotherapy failure is defined as disease progression or intolerable toxicity during treatment or within 3 months after the last dose; If patients cannot receive the above treatment for economic reasons, those whose benefits outweigh the risks of inclusion in the study can be enrolled.
4. Subjects with positive CEA (IHC score 3+) in tumor tissue samples (paraffin sections or fresh tissue specimens or puncture biopsy samples) within 3 months before screening; If the immunohistochemical results of the tumor samples are more than 3 months from the time of screening, the patient needs to re-biopsy; If the tumor specimens are not available or the amount is too small for immunohistochemical detection of CEA, the CEA positive can be confirmed by re-staining of previous tissue specimens, and the peripheral blood serum CEA≥2.0×ULN can be included in the group.
5. Have at least one evaluable target lesion according to RECIST 1.1 criteria;
6. Colorectal cancer, esophageal cancer, non-small cell lung cancer, breast cancer, stomach cancer, cholangiocarcinoma ECOG 0 ~ 1 score, pancreatic cancer ECOG 0 ~ 2 score;
7. Expected survival time is more than 12 weeks;
8. No serious mental disorders;
9. Unless otherwise stated, the subject's vital organ functions shall meet the following conditions:

   1. Blood routine: white blood cells > 3.5×109/L, neutrophils > 1.8×109/L, lymphocytes > 0.5 ×109/L, platelet > 80×109/L, hemoglobin > 90g/L;
   2. Cardiac function: Echocardiography indicated cardiac ejection fraction ≥50%, and no obvious abnormality was found in electrocardiogram;
   3. Renal function: serum creatinine ≤2.0×ULN;
   4. Liver function: ALT and AST≤3.0×ULN (patients with liver tumor infiltration can be relaxed to ≤5.0 ×ULN);
   5. Total bilirubin ≤2.0×ULN (Gilbert syndrome ≤3.0×ULN; The patients with liver tumor infiltration can be enlarged to ≤5.0×ULN);
   6. Blood oxygen saturation in non-oxygen state > 92%.
10. Have the criteria for simple or intravenous blood collection, and no other contraindications for cell collection;
11. The subject agrees to use a reliable and effective method of contraception (excluding safe period contraception) for 1 year from signing the informed consent to receiving the C-13-60 cell infusion. Including but not limited to: abstinence, can inhibit ovulation implantable progesterone contraceptive; Intrauterine device (IUD); Intrauterine hormone release system; Spousal vasectomy; Combined hormonal contraceptives (oral, vaginal, and transdermal) that inhibit ovulation; Progesterone contraceptives (oral or injectable) that inhibit ovulation; Male subjects who have sex with fertile women must consent to the use of a barrier method of contraception (e.g., condom plus spermicidal foam/gel/film/emulsion/suppository). At the same time, the subject should promise not to donate eggs (egg cells, oocytes) or sperm for assisted reproduction within 1 year after the cell infusion.
12. The patient or his/her guardian agrees to participate in the clinical trial and signs the ICF, indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. People who have received CAR-T therapy or other gene-modified cell therapy;
2. Patients with BMS with clinical symptoms or lesions located in key parts of the brain at the time of screening, patients with BMS without clinical symptoms or lesions located in non-critical parts of the brain should be evaluated by researchers or specialists to gain more than the risk.
3. Received any of the following medications or treatments before screening:

   1. Received other investigational drugs or treatments that are not on the market within 4 weeks prior to screening;
   2. Received live attenuated vaccine within 4 weeks prior to screening;
   3. Received radioactive iodine-125 particle implantation within 8 weeks prior to screening;
4. Received the following drugs or treatments before apheresis:

   1. received the equivalent of &gt within 2 weeks prior to apheresis; 10mg/ day of prednisone for systemic steroids, except inhaled steroids;
   2. Received anti-PD-1 / PD-L1 monoclonal antibody treatment within 4 weeks before apheresis; Received chemotherapy, targeted therapy, or other investigational agents within 2 weeks of preapheresis or at least 5 drug half-lives (whichever is shorter);
5. There is an active or uncontrolled infection that requires systemic treatment within 1 week prior to screening;
6. Subjects with intestinal obstruction, active gastrointestinal bleeding, history of massive gastrointestinal bleeding within 3 months, severe gastroduodenal ulcer, severe ulcerative colitis and other severe intestinal inflammation;
7. History of severe respiratory disease;
8. There are a large number of serous effusions that cannot be controlled by treatment (such as pleural effusions, abdominal effusions and pericardial effusions);
9. Have any of the following heart conditions:

   1. New York Heart Association (NYHA) Stage III or IV congestive heart failure;
   2. Had myocardial infarction or coronary artery bypass grafting (CABG) within ≤6 months before enrollment;
   3. A history of clinically significant ventricular arrhythmia, or unexplained syncope (other than those caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy.
10. Known to have active or uncontrolled autoimmune diseases that require treatment with immunosuppressants, including biologics, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, systemic vasculitis, etc.;
11. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA test greater than the normal range; Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA detection greater than the normal range; Human immunodeficiency virus (HIV) antibody positive; Syphilis positive; Cytomegalovirus (CMV) DNA test positive;
12. At the time of screening, subjects had venous embolism events (e.g., pulmonary embolism) and required anticoagulant therapy;
13. Other uncured malignant tumors within the past 3 years or at the same time, except cervical carcinoma in situ and skin basal cell carcinoma;
14. Women who are pregnant or nursing, and male or female subjects who plan to have a child within 1 year after receiving C-13-60 cell transfusion;
15. Circumstances deemed unsuitable for participation in the study by other researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the dose range and DLT of C-13-60 cells for CEA positive advanced malignant solid tumors [Safety and Tolerability] | 1 month
  The incidence of adverse events (TEAE) after treatment; Incidence of treatment-related adverse events; Adverse evens of Special Interest (AESI);
To obtain the maximum tolerable dose of C-13-60 cells [Safety and Tolerability] | 1month
  Incidence and number of dose-limiting toxicity (DLT) cases，Dose-limiting toxicity after CAR-T cell infusion

SECONDARY OUTCOMES:
Disease control rate (DCR) within 3 months after infusion of C-13-60 cell preparation[Effectiveness] | 3 months
  Disease control rate: The proportion of subjects who achieved complete response (CR), partial response (PR), stable disease (SD) after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Area under the curve (AUCS) of C-13-60 cell [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
Maximum concentration (CMAX) of C-13-60 cell [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CEA CAR-T cells expanded in peripheral blood
Maximum time (TMAX) of C-13-60 cell[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
The content of CEA in peripheral blood after infusion of C-13-60 cell [Cell dynamics] | 3 months
  The concentration of serum CEA in peripheral blood was detected by ELISA at the visit points specified in the research protocol

OTHER OUTCOMES:
Objective response rate (ORR) of C-13-60 cell treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  Objective response rate includes：The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of C-13-60 cell treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of C-13-60 cell treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS) of C-13-60 cell treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause (Assessed by investigators based on RECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, M.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Weijia Fang, M.D, Principal Investigator — Zhejiang University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang